CLINICAL TRIAL: NCT01478607
Title: A Randomized, Controlled, Long-term Safety Study Evaluating the Effect of Repeated Applications of QUTENZATM Plus Standard of Care Versus Standard of Care Alone in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: A Study to Evaluate the Long-term Safety of Repeated QUTENZA Administration for Treatment of Pain Caused by Nerve Damage in Diabetic Patients
Acronym: PACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E05-CL-3002; 2009-016458-42 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Painful Diabetic Peripheral Neuropathy (PDPN)
Keywords: Painful Diabetic Peripheral Neuropathy; Qutenza
MeSH Terms: interventions — Capsaicin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Qutenza 30 minutes + SOC (Experimental)
  Interventions: Drug: QUTENZA
- 2. Qutenza 60 minutes + SOC (Experimental)
  Interventions: Drug: QUTENZA
- 3. SOC (No Intervention): Subjects randomized to this group will receive treatment optimized for them on an individual basis. The investigator will be free to provide whatever pharmacological or other treatment is considered optimal for management of the subject's pain.

INTERVENTIONS:
Drug: QUTENZA — A Qutenza (8% capsaicin) patch will be applied to identified painful areas for 30 minutes (Arm 1) or 60 minutes (Arm 2).
  Other Names: Capsaisin
  Arms: 1. Qutenza 30 minutes + SOC; 2. Qutenza 60 minutes + SOC

SUMMARY:
The purpose of the study is to assess the safety of repeated applications of QUTENZA in reducing pain intensity in subjects who have peripheral neuropathic pain due to diabetes.

DETAILED DESCRIPTION:
Patients will be divided into 3 groups of approximately equal size. In the first group, patients will receive a QUTENZA patch applied for 30 minutes to the feet; in the second group, patients will receive a QUTENZA patch applied for 60 minutes to the feet. In both these groups patients will also continue to receive their normal treatment (Standard of Care (SOC)) for their peripheral neuropathic pain (PNP) and may receive further QUTENZA patch applications in the same way during the study. The third group will not receive a QUTENZA patch but will continue to receive their normal treatment for their neuropathic pain (SOC). Subjects will be involved in the study for up to 15 months and will have to visit the clinic at least 9 times.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of painful, distal, symmetrical, sensorimotor polyneuropathy which is due to diabetes
* Stable glycemic control for at least 6 months prior to screening visit
* Average Numeric Pain Rating Scale (NPRS) score over the last 24 hours of >4 at the screening and the baseline visit

Exclusion Criteria:

* Primary pain associated with PDPN in the ankles or above
* Pain that could not be clearly differentiated from, or conditions that might interfere with, the assessment of PDPN
* Significant pain (moderate or above) of an etiology other than PDPN, that may interfere with judging PDPN-related pain
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test at enrollment and must agree to maintain highly effective birth control during the study.
* Hypersensitivity to capsaicin (i.e., chili peppers or over-the-counter [OTC] capsaicin products), any QUTENZA excipients, Eutectic Mixture of Local Anesthetics( EMLA) ingredients or adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Percentage change in health related quality of life (HRQOL) total score as assessed by the disease specific Norfolk scale | Baseline till endpoint (discontinuation or End of Study visit) (up to 64 weeks)

SECONDARY OUTCOMES:
Neurological function as assessed by the Utah Early Neuropathy Scale (UENS) and sensory testing | Baseline till End of Study (up to 64 weeks)
  Physicians measuring neurological function will be blinded to treatment
Tolerability of patch application by dermal assessment | Screening till Last visit when QUTENZA patch is applied (up to 53 weeks)
Tolerability of patch application by "pain now" Numeric Pain Rating Scale (NPRS) scores after patch application | Baseline till Last visit when QUTENZA patch is applied (up to 52 weeks)
  Assessed within 15 minutes and 60 minutes after patch removal.
Tolerability of patch application by rescue medication use | Days 1 through 5 after each patch application
Adverse Events and serious adverse Events | Screening visit through End of study visit (up to 65 weeks)
Vital Signs (heart rate and blood pressure) | Screening visit through End of study visit (up to 65 weeks)
  In case of patch application to be performed within 15 minutes before topical anesthetic application and within 15 minutes after patch removal.
Laboratory Analyses | Screening visit through End of study visit (up to 65 weeks)
  The tests performed at the screening visit will include Hematology: Red Blood Cell Count, White Blood Cell Count, Lymphocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Hemoglobin, Hematocrit and Platelets. Biochemistry: Aspartate Aminotransferase (AST) and/or Alanine Aminotransferase (ALT), Alkaline Phosphatase, Sodium, Potassium, Blood Urea Nitrogen (BUN), Creatinine and Lipid profile. Subsequent HbA1c and lipid profile follow-up will be done at bi-monthly visits. The other tests will be performed if clinically indicated.
Intensity of neuropathic pain using "average pain" NPRS scores | Screening visit through End of study visit (up to 65 weeks)
  Question 5 of Brief Pain Inventory-Diabetic Neuropathy (BPI-DN)
Brief Pain Inventory (BPI) pain severity index and pain interference index | Screening visit through End of study visit (up to 65 weeks)
Patient Global Impression of Change | After each patch re-application, from first patch re-application through End of Study visit (up to 56 weeks)
Generic HRQOL measured by European Quality of Life - 5 Dimensions (EQ-5D) questionnaire | After each patch application, from first patch application through End of Study (up to 64 weeks)
Treatment satisfaction using the Self-Assessment of Treatment (SAT) questionnaire at week 12/End Of Study visit | End of Study (up to 65 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Clinical Study Manager, Study Director — Astellas Pharma Europe B.V.
Locations (64):
- Site: 601, Bonheiden, Belgium
- Czechia (9):
  - Site: 903, Beroun
  - Site: 910, Brno
  - Site: 908, Choceň
  - Site: 911, Litoměřice
  - Site: 906, Ostrava
  - Site: 904, Polička
  - Site: 901, Prague
  - Site: 902, Přerov
  - Site: 909, Rychnov nad Kněžnou
- France (4):
  - Site: 207, Bron
  - Site: 202, Paris
  - Site: 201, Pierre-Bénite
  - Site: 206, Toulouse
- Germany (9):
  - Site: 508, Chiemsee
  - Site: 509, Cologne
  - Site: 502, Dresden
  - Site: 501, Falkensee
  - Site: 514, Frankfurt
  - Site: 507, Hamburg
  - Site: 505, Leipzig
  - Site: 506, Münster
  - Site: 512, Wangen
- Italy (2):
  - Site: 404, Milan
  - Site: 401, Roma
- Site: 651, Utrecht, Netherlands
- Poland (11):
  - Site: 965, Bialystok
  - Site: 961, Bydgoszcz
  - Site: 957, Elblag
  - Site: 958, Gdynia
  - Site: 954, Katowice
  - Site: 964, Krakow
  - Site: 951, Lodz
  - Site: 966, Lubin
  - Site: 953, Poznan
  - Site: 959, Torun
  - Site: 960, Warsaw
- Russia (9):
  - Site: 714, Kemerovo
  - Site: 703, Saint Petersburg
  - Site: 716, Saint Petersburg
  - Site: 704, Saint Petersburg
  - Site: 706, Saint Petersburg
  - Site: 708, Samara
  - Site: 709, Saratov
  - Site: 713, Tomsk
  - Site: 711, Yaroslavl
- Spain (3):
  - Site: 303, Valencia
  - Site: 304, Valencia
  - Site: 305, Valladolid
- Ukraine (11):
  - Site: 808, Chernihiv
  - Site: 803, Kharkiv
  - Site: 812, Kvuv
  - Site: 805, Kyiv
  - Site: 807, Kyiv
  - Site: 806, Kyiv
  - Site: 810, Lviv
  - Site: 802, Mykolayiv
  - Site: 801, Odesa
  - Site: 813, Vinnitsa
  - Site: 815, Zaporizhzhya
- United Kingdom (4):
  - Site: 102, Chorley
  - Site: 103, Liverpool
  - Site: 104, Poole
  - Site: 101, Rugby

REFERENCES:
- [Derived] Vinik AI, Perrot S, Vinik EJ, Pazdera L, Jacobs H, Stoker M, Long SK, Snijder RJ, van der Stoep M, Ortega E, Katz N. Capsaicin 8% patch repeat treatment plus standard of care (SOC) versus SOC alone in painful diabetic peripheral neuropathy: a randomised, 52-week, open-label, safety study. BMC Neurol. 2016 Dec 6;16(1):251. doi: 10.1186/s12883-016-0752-7. PMID 27919222
- See also: Link to results on EudraCT — https://www.clinicaltrialsregister.eu/ctr-search/trial/2009-016458-42/results
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/study.aspx?ID=E05-CL-3002